CLINICAL TRIAL: NCT05056753
Title: Amerlioration of Opioid Withdrawal-Induced Anxiety and Craving With Heterodyned Whole-Body Vibration (HWBV)
Brief Title: Heterodyned Whole-Body Vibration in Treatment of Opioid Withdrawal-Induced Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PhotoPharmics, Inc. (Industry)
Collaborators: Brigham Young University (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CT2101; R41DA053083-01A1 (NIH)
Record Dates: First submitted 2021-06-25; First posted 2021-09-27 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-10

CONDITIONS: Opioid-use Disorder
Keywords: Opioid-use Disorder; Addiction, Opioid
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Intervention Model Description: This is a 4-week, randomized, double-blind, controlled, parallel group study with 5 visits; at screening/baseline, and weeks 1-4 and daily visits to the treatment clinic, with blinded evaluation of efficacy and safety assessments.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants will spend approx 30 min/day for 5 days/week in HWBV testing for the 4-week treatment period at the treatment clinic. Eligible participants who consent to the study are screened and randomized to either the active or control group, using the vibration device with controller that has 2 unmarked presets as to which treatment protocol they represent (HWBV or monotonic vibration). Neither the study coordinator, technician, nor site investigator will know which setting is the active or control. The device technician (blinded to the treatment hypothesis) will help participants set up the device and provide assistance. To avoid unblinding, device technician will be segregated from all study personnel and data. He/she will also be instructed not to comment to the patients on any aspects of the device and defer study related questions to the study staff. A blinded coordinator / staff member will conduct study assessments at baseline, weeks 1, 2, 3, and 4, visits.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Investigational Device (Active Comparator): The HWBV chair consists of a custom-made saddle-seat type of chair. The vibration actuators are embedded into the underside design of the chair. The base contains two vibrators, one for each side of the chair, and the chair is split in half vertically so that the vibrating actuators are able to send a harmonic vibration at alternating frequencies, upwards through each side of the chair. The HWBV system is considered a non-significant and non-substantial risk device.
  Interventions: Device: HWBV chair
- Control Device (Sham Comparator): The Control device is identical in construction to the Active device. The vibration mode, however, is a significantly different setting than that used by the Active version, so that the mechanoreceptors in the cervical spine are not effectively stimulated.
  Interventions: Device: HWBV chair

INTERVENTIONS:
Device: HWBV chair — vibration-actuated, saddle-seat type stool

SUMMARY:
In this randomized, double-blind, controlled, parallel group study (conducted over 12-months), enrollment is expected of up to 60 subjects (30 men and 30 women) ages 18+ who are currently going through withdrawal of OUD and being treated at local substance abuse clinics. The study visits will include screening, baseline, Weeks 1, 2, 3, and 4, with both safety and efficacy assessments.

DETAILED DESCRIPTION:
Approximate time commitment is 30 minutes / day, for 5 days / week, in testing effects of specialized 'massage' chair for a period of 4 weeks (up to total 20 treatment periods). Only about 20 minutes time is in the test chair, and the rest is setup time and completing questionnaires.

* Upon arrival to the clinic for treatment, some short questions are asked.
* Participant is seated in a HWBV chair device.
* A clip is attached to one finger to track heart rate and skin response to the treatment.
* After relaxing for about 5 minutes, the HWBV chair actuated for 10 minutes.
* The finger attachment is disconnected.
* Post-treatment, some more survey questions conclude the session.

ELIGIBILITY:
Inclusion Criteria:

* Minimum age of 18 (female and male)
* Confirmed diagnosis of opioid use disorder and deemed appropriate to participate in this study as referred by the medial director of a local outpatient treatment clinic for OUD
* Concurrent craving for drug
* In otherwise good physical health
* Access to a phone (communication device) and willingness to communicate with study staff
* Ability to understand and provide informed consent in English

Exclusion Criteria:

* Inability to provide verifiable contact information or unwillingness to assist with follow-up
* Unwilling to allow potential access to medical, drug treatment records or criminal history or criminal activity records that in the opinion of the site investigator would interfere with the conduct of the study
* History of violence or violent, erratic behavior that would indicate a risk to other participants, study staff or to the participant her/himself
* Psychoses, major depression, bipolar disorder, or other mental disorder that in the opinion of the site investigator, would interfere with the participant's ability to participate in the study
* A score of > 2 on the Beck Depression Inventory-II (BDI-II) [Suicidality]
* A score of < 6 on the Clinical Opiate Withdrawal Scale, which indicates mild opiate withdrawal symptoms
* Prior history of severe brain injury or seizures
* Prone to fainting
* Suffering from a recent injury from which they are still recovering or needing medications for recovery
* Not have used opiates within the last 24 hours or longer than the past 60 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2022-01-20 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-07-30 (Actual)

PRIMARY OUTCOMES:
Hamilton Anxiety Rating Scale (HAM-A) | 4 weeks
  The Hamilton Anxiety Rating Scale (HAM-A) measures severity of anxiety, with 14 domains and is administered by a clinician. Severity is rated from 0 - 4 on each question, with a total possible of 56 points. A higher score is reflects worse severity

SECONDARY OUTCOMES:
Clinical Opiate Withdrawal Scale (COWS) | 4 weeks
  The Clinical Opiate Withdrawal Scale (COWS) is an 11-item scale designed to rate common signs and symptoms of opiate withdrawal to show overall severity of addiction. Each question ranks severity from 0-4 or 5, depending on the question. A higher score indicates greater severity. The COWS to be administered by a clinician

OTHER OUTCOMES:
Physiologic Assessment: Galvanic skin response (GSR) | 4 weeks
  Physiologic measures of Galvanic skin response (GSR), will be measured during the 5-minute pre-, the 10-minute seated vibration session, and 5-minute post-vibration in the chair (device technician will then remove the finger plethysmograph).
Physiologic Assessment: Heart rate (HR) | 4 weeks
  Physiologic measures of heart rate (HR), will be measured during the 5-minute pre-, the 10-minute seated vibration session, and 5-minute post-vibration in the chair (device technician will then remove the finger plethysmograph).
Physiologic Assessment: Heart rate variability (HRV) | 4 weeks
  Physiologic measures of heart rate variability (HRV), will be measured during the 5-minute pre-, the 10-minute seated vibration session, and 5-minute post-vibration in the chair (device technician will then remove the finger plethysmograph).

CONTACTS AND LOCATIONS:
Locations (1):
- Migraine and Neuro Rehab Clinic, Provo, Utah, United States

IPD SHARING:
Plan to Share IPD: Yes
In addition to submitting the study design and results to www.clinicaltrials.gov, the final results of the study will be published in a peer-reviewed journal after the generation of the clinical study report. Subsequent to publication, PhotoPharmics and Brigham Young University intend to make the data available to qualified researchers for collaboration. The general results of the trial may also be made available to study participants during a webinar.